CLINICAL TRIAL: NCT01334086
Title: A Phase II Open Label Study of Aprepitant as Antiemetic Prophylaxis in Patients With Acute Myeloid Leukemia Undergoing Induction Chemotherapy
Brief Title: Aprepitant as Antiemetic Prophylaxis in Patients With Acute Myeloid Leukemia Undergoing Induction Chemotherapy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: AML-11-001
Record Dates: First submitted 2011-03-25; First posted 2011-04-12 (Estimated); Results first posted 2021-05-11 (Actual); Last update posted 2021-11-22 (Actual); Status verified 2021-04

CONDITIONS: Acute Myeloid Leukemia
Keywords: AML
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — Aprepitant

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Aprepitant (Experimental)
  Interventions: Drug: Aprepitant

INTERVENTIONS:
Drug: Aprepitant — Oral aprepitant will be given to the participant on Days 1-5 of standard induction treatment. A dose of 125 mg will be given on Day 1 and 80 mg will be given on Days 2-5.
  Other Names: Emend

SUMMARY:
Chemotherapy induced nausea and vomiting (CINV) is a major adverse effect of chemotherapy. This study is determining the incidence of vomiting/retching of the standard induction chemotherapy regimen for patients with acute myeloid leukemia (AML) who are also receiving an antiemetic known as aprepitant.

The standard frontline chemotherapy for patients with AML consists of cytarabine given as a 7 day continuous infusion plus 3 days of an anthracycline, most commonly daunorubicin, on days 1-3. This is known as the 3+7 regimen. Antiemetic treatments are usually given to patients for nausea and vomiting. Granisetron (a 5-HT3 receptor antagonist) is used on the 3 daunorubicin days and other antiemetics can be used for breakthrough nausea/vomiting.

This study will test that the prophylactic use of aprepitant, in addition to the standard antiemetic regimen used at Princess Margaret Hospital (PMH), will reduce the incidence of delayed onset vomiting/retching by Day 5 in AML patients receiving the standard 3+7 regimen, compared to retrospective data using this regimen.

ELIGIBILITY:
Inclusion Criteria:

* Acute myeloid leukemia (AML), any subtype including acute promyelocytic leukemia (APL). Patients with either de novo or secondary AML are eligible.
* No prior AML induction chemotherapy.
* Due to receive standard 3+7 induction chemotherapy using daunorubicin on Days 1-3, plus cytarabine continuous infusion daily on Days 1-7.
* Age 18 and over.
* Serum bilirubin < or = 1.5 times the upper limit of normal (ULN).
* Serum aspartate aminotransferase and alanine aminotransferase < or = 2.5 times the ULN.
* Serum creatinine < 200 umol/L

Exclusion Criteria:

* Uncontrolled nausea or vomiting within 48 hours prior to start of induction therapy. Grade 0-1 nausea is permitted at the start of induction.
* Known hypersensitivity to granisetron or aprepitant.
* Patients currently receiving treatment with strong CYP3A4 inhibitors or substrates and treatment cannot be either discontinued or switched to a different medication prior to starting study drug.
* Not able to swallow or absorb oral medications.
* Documented active central nervous system (CNS) leukemia or recent CNS hemorrhage.
* Concomitant use of:

  1. Other investigational agents during induction therapy
  2. Radiotherapy during, or one month prior to, induction therapy
  3. Systemic corticosteroids
  4. Other chemotherapy agents on Days 1-8
* Pregnant or breast feeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2011-09; Primary Completion 2013-08 (Actual); Study Completion 2013-08-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joseph M Brandwein, MD, FRCPC, Principal Investigator — University Health Network - Princess Margaret Hospital
Locations (1):
- Princess Margaret Hospital, Toronto, Ontario, Canada

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Aprepitant
Started | 41
Completed | 41
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Aprepitant
Number analyzed (Participants) | 41
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 26
  >=65 years | 15
Age, Continuous [Median (Full Range); unit: years] | 56 [22 to 78]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18
  Male | 23
Region of Enrollment [Number; unit: participants]
  Canada | 41

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Incidence of Vomiting/Retching From Day 1 Through End of Day 5
Description: Cumulative incidence will be determined by the patient self-assessment form, supplemented by the nursing inpatient records.
Time Frame: Day 1 through end of Day 5
Measure: Number; unit: percentage of particpants
Arm/Group | Aprepitant
Number analyzed (Participants) | 38
percentage of particpants | 26.3

2. Secondary Outcome: Presence of Nausea Per Day, on Days 1-8.
Time Frame: Days 1 to 8
Reporting Status: Not Posted

3. Secondary Outcome: Daily Number of Vomiting or Retching Incidents From Days 1-8
Description: This will be determined by both self-assessment form which will be filled out by the patient on a daily basis, and review of the nursing inpatient records.
Time Frame: Days 1 to 8
Measure: Number; unit: incidents
Arm/Group | Aprepitant
Number analyzed (Participants) | 38
incidents
  Day 1 | 7
  Day 2 | 11
  Day 3 | 16
  Day 4 | 13
  Day 5 | 13
  Day 6 | 24
  Day 7 | 13
  Day 8 | 11

4. Secondary Outcome: Percentage of Participants Experiencing Vomiting or Retching From Days 1-8.
Description: as for outcome 3
Time Frame: Days 1 to 8
Measure: Number; unit: percentage of particpants
Arm/Group | Aprepitant
Number analyzed (Participants) | 38
percentage of particpants | 34.2

5. Secondary Outcome: Percentage of Patients Experiencing Nausea From Days 1-8.
Time Frame: Days 1 to 8
Measure: Number; unit: percentage of particpants
Arm/Group | Aprepitant
Number analyzed (Participants) | 38
percentage of particpants | 68.4

6. Secondary Outcome: Percentage of Patients' Use of Supplemental Anti-emetics as Determined by the Total Number of Doses Per Day and in Total, From Days 1-8.
Time Frame: Days 1 to 8
Measure: Number; unit: % of pts receiving breakthrough
Arm/Group | Aprepitant
Number analyzed (Participants) | 41
% of pts receiving breakthrough
  Day 1 | 18
  Day 2 | 29
  Day 3 | 39
  Day 4 | 58
  Day 5 | 65
  Day 6 | 75
  Day 7 | 68
  Day 8 | 53

7. Secondary Outcome: To Evaluate the Tolerance of Aprepitant by Documenting All Toxicities on Days 1-8 and All Unexpected Serious Adverse Events up to Day 30.
Time Frame: Days 1 to 8
Reporting Status: Not Posted

8. Secondary Outcome: Severity of Nausea Per Day, on Days 1-8.
Time Frame: Days 1 to 8
Reporting Status: Not Posted

ADVERSE EVENTS:
Arm/Group | Aprepitant
Serious Adverse Events (participants affected / at risk) | 2/41
Other Adverse Events (participants affected / at risk) | 40/41
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Aprepitant (N=41)
Vomitting (Gastrointestinal disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Aprepitant (N=41)
ABDOMINAL DISTENSION (Gastrointestinal disorders) | 2 (2)
ABDOMINAL PAIN (Gastrointestinal disorders) | 3 (3)
ANEMIA (Blood and lymphatic system disorders) | 2 (2)
ANOREXIA (Metabolism and nutrition disorders) | 13 (13)
ANXIETY (Psychiatric disorders) | 5 (5)
BACK PAIN (Musculoskeletal and connective tissue disorders) | 3 (3)
BLURRED VISION (Eye disorders) | 4 (4)
BRUISING (Injury, poisoning and procedural complications) | 3 (3)
CHILLS (General disorders) | 9 (10)
CONSTIPATION (Gastrointestinal disorders) | 2 (2)
COUGH (Respiratory, thoracic and mediastinal disorders) | 6 (6)
DEPRESSION (Psychiatric disorders) | 2 (2)
DIARRHEA (Gastrointestinal disorders) | 18 (19)
DIZZINESS (Nervous system disorders) | 10 (10)
DRY MOUTH (Gastrointestinal disorders) | 3 (3)
DYSGEUSIA (Nervous system disorders) | 4 (4)
DYSPEPSIA (Gastrointestinal disorders) | 5 (5)
EPISTAXIS (Respiratory, thoracic and mediastinal disorders) | 6 (6)
EYE PAIN (Eye disorders) | 2 (2)
FATIGUE (General disorders) | 10 (10)
FEBRILE NEUTROPENIA (Blood and lymphatic system disorders) | 19 (19)
FEVER (General disorders) | 4 (4)
FLUSHING (Vascular disorders) | 3 (3)
HEADACHE (Nervous system disorders) | 16 (16)
HEMORRHOIDS (Gastrointestinal disorders) | 3 (3)
HYPERHIDROSIS (Skin and subcutaneous tissue disorders) | 4 (4)
HYPOKALEMIA (Metabolism and nutrition disorders) | 6 (6)
HYPOPHOSPHATEMIA (Metabolism and nutrition disorders) | 3 (3)
HYPOTENSION (Vascular disorders) | 13 (14)
HYPOXIA (Respiratory, thoracic and mediastinal disorders) | 2 (2)
INSOMNIA (Psychiatric disorders) | 4 (4)
MUCOSITIS ORAL (Gastrointestinal disorders) | 19 (21)
NAUSEA (Gastrointestinal disorders) | 25 (27)
NECK PAIN (Musculoskeletal and connective tissue disorders) | 3 (3)
DYSOSMIA (General disorders) | 2 (2)
NEUTROPHIL COUNT DECREASED (Investigations) | 4 (5)
ORAL HEMORRHAGE (Gastrointestinal disorders) | 2 (2)
ORAL PAIN (Gastrointestinal disorders) | 4 (4)
PAIN (General disorders) | 3 (3)
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 5 (5)
PARESTHESIA (Nervous system disorders) | 4 (4)
PLATELET COUNT DECREASED (Investigations) | 2 (2)
PRODUCTIVE COUGH (Respiratory, thoracic and mediastinal disorders) | 4 (4)
PRURITUS (Skin and subcutaneous tissue disorders) | 10 (11)
RASH ACNEIFORM (Skin and subcutaneous tissue disorders) | 9 (9)
RASH MACULO-PAPULAR (Skin and subcutaneous tissue disorders) | 9 (10)
SEPSIS (Infections and infestations) | 2 (2)
SINUS BRADYCARDIA (Cardiac disorders) | 3 (3)
SKIN INFECTION (Infections and infestations) | 5 (6)
SKIN ULCERATION (Skin and subcutaneous tissue disorders) | 2 (5)
SORE THROAT (Respiratory, thoracic and mediastinal disorders) | 3 (3)
STOMACH PAIN (Gastrointestinal disorders) | 2 (2)
URINARY INCONTINENCE (Renal and urinary disorders) | 2 (2)
VOMITING (Gastrointestinal disorders) | 4 (4)
EDEMA LIMBS (General disorders) | 8 (10)
LUNG INFECTION (Infections and infestations) | 5 (5)
LOCALIZED EDEMA (General disorders) | 2 (2)
GENERALIZED MUSCLE WEAKNESS (Musculoskeletal and connective tissue disorders) | 4 (4)
PAPULOPUSTULAR RASH (Infections and infestations) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No